CLINICAL TRIAL: NCT04962828
Title: The Effect Of An Inter Disciplinary Approach On Vocabulary Development in Children With Hearing Impairment; A Randomized Control Trial
Brief Title: Inter Disciplinary Approach to Vocabulary Development in Hearing Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00973
Record Dates: First submitted 2021-07-10; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Hearing Impaired Children
Keywords: Hearing Impairment; Language Intervention; Interdisciplinary working
MeSH Terms: conditions — Hearing Loss | interventions — Communication Methods, Total; Language Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaboration group (Experimental): This group of children will have targets and vocabulary that has been designed collaboratively and then the therapist and teacher both reinforce the vocabulary during the week
  Interventions: Other: Vocabulary based intervention - Collaborative
- Non-collaborative group (Active Comparator): This group of children will have targets and vocabulary that has been designed collaboratively but they will only be practiced with the therapist during the week
  Interventions: Other: Vocabulary based intervention- Non Collaborative

INTERVENTIONS:
Other: Vocabulary based intervention- Non Collaborative — List of 10 words functional words Therapy 3 times a week for 20 minutes Duration = 9 weeks Only with SLP
  Other Names: Language Intervention; Language Intervention for Hearing Impairment; Total Communication
  Arms: Non-collaborative group
Other: Vocabulary based intervention - Collaborative — List of 10 words functional words Therapy 3 times a week for 20 minutes Duration = 9 weeks With SLP and to be reinforced by teachers in class over the week
  Other Names: Language Therapy; Inter-disciplinary working
  Arms: Collaboration group

SUMMARY:
The research aims to address to address the role of interdisciplinary working between professionals in the field of speech and language pathology/therapy. There is considerable evidence to state that when professionals work in collaboration with each other on particular goals that the outcomes are more favorable, functional and beneficial for the child.

DETAILED DESCRIPTION:
The aim of the current research is to devise a joint interventional program between the speech and language pathologist and teachers in order to support their comprehension and expression of functional vocabulary. This study was devised as there is a gap in collaborative working by professionals in Pakistan. Often therapy is provided through a medical model of taking the child outside the class for one to one sessions. There is lack of lack of collaborative goal planning. This is particularly true for children who are in hearing impairment centres.

In Pakistan, the prevalence of all hearing loss in rural Pakistan has been estimated to be 7.9%, in a general population setting. The high prevalence rates are a source of concern. The impact of hearing impairment manifests itself in many ways. As is evident from the studies carried out on the impact of hearing impairment on vocabulary skills and speech-language and communication difficulties in general of children and adolescents, that these difficulties if not identified in a timely manner will affect later schooling and educational attainment. Vocabulary knowledge is a key predictor of reading comprehension, which is essential for academic progress.

In the field of early intervention and early childhood special education caregiver involvement has been documented as important. Speech, language and communication needs (SLCN) are prevalent among primary school-aged children. Collaboration between speech and language therapists (SLTs) and teachers is beneficial for supporting children's communication skills. Findings from an Australian study suggests that change to service delivery needs to be considered at an individual, interpersonal and organizational level to enable better outcomes for children with SLCN and increased support for their families and the professionals who work with them.

Hence, timely identification and management plays a pivotal role. It is critical that therapy is provided in a manner as to generalize learnt skills. Research described speech therapy services as largely happening outside of the classroom such as removing individuals or small groups from the classroom for intervention sessions ('pull out') or that involve the speech-language pathologist indirectly affecting the child's educational program by providing modeling or coaching to relevant educators in the use of strategies to promote specific skills ('consultation').

There is no denying that collaborative working is essential. A study comparing improvement on a specific study measure designed on selected vocabulary in 12 classrooms with 3 conditions: (1) Pull-out - 50-minute group or one to one sessions for twelve weeks. (2) Classroom-based - Weekly 40-minute lessons for 12 weeks (3) Collaborative - Weekly 40-minute SLP-teacher planned and team taught lessons for 12 weeks. The results suggested evidence for the benefits of collaborative working such as the ability to discuss, design and plan between the teacher and SLP, resulting in greater outcomes and facilitating generalization of the activities in students who require it the most. The study sheds light on the need for such collaboration and provides evidence sums for further research to address similar outcomes in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impaired children from 6 to 11 years of age who have severe unilateral or bilateral hearing loss from birth and for whom Urdu has their first language. There hearing age is at least one year. Their parents were not hearing impaired. Children used hearing aids. Unilateral & bilateral hearing impaired children were equally distributed.

Exclusion Criteria:

* Children who did not present with HI as their main diagnosis or may have other co-morbid conditions.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-07-26 (Estimated); Study Completion 2021-07-26 (Estimated)

PRIMARY OUTCOMES:
Vocabulary List | 9th week
  There will be 10 functional words that will be designed post collaboration with the teachers. The list will accommodate 6 Ling sounds and will be implemented with both groups. The participants will be tested on the list pre-intervention and post intervention. Scoring will be based on binary responses such as correct and incorrect responses. Any further responses will be addressed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Butt, PhD, Principal Investigator — Riphah International University
Locations (1):
- Aghosh Special Children's School, Kharian, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Background] Mathers C, Smith A, Concha M. Global Burden Of Hearing Loss In The Year 2000. Global Burden Of Disease. 2000;18(4):1-30.
- [Background] McGregor KK, Oleson J, Bahnsen A, Duff D. Children with developmental language impairment have vocabulary deficits characterized by limited breadth and depth. Int J Lang Commun Disord. 2013 May-Jun;48(3):307-19. doi: 10.1111/1460-6984.12008. Epub 2013 Feb 25. PMID 23650887
- [Background] Suleman S, Mcfarlane La, Pollock K, Schneider P, Leroy C, Skoczylas M. Collaboration: More Than
- [Background] Ebbels SH, McCartney E, Slonims V, Dockrell JE, Norbury CF. Evidence-based pathways to intervention for children with language disorders. Int J Lang Commun Disord. 2019 Jan;54(1):3-19. doi: 10.1111/1460-6984.12387. Epub 2018 Apr 25. PMID 29696726
- [Background] Wilson L, McneillBc, Gillon Gt. Understanding The Effectiveness Of Student Speech-Language Pathologists And Student Teachers Co-Working During Inter-Professional School Placements. Child Language Teaching And Therapy. 2019 Jun;35(2):125-43.( 7)
- [Background] Lowe H, Henry L, Joffe VL. The Effectiveness of Classroom Vocabulary Intervention for Adolescents With Language Disorder. J Speech Lang Hear Res. 2019 Aug 15;62(8):2829-2846. doi: 10.1044/2019_JSLHR-L-18-0337. Epub 2019 Jul 24. PMID 31339808
- [Background] Glover A, Mccormack J, Smith-Tamaray M. Collaboration Between Teachers And Speech And Language Therapists: Services For Primary School Children With Speech, Language And Communication Needs. Child Language Teaching And Therapy. 2015 Oct;31(3):363-82.
- [Background] Murray E, McCabe P, Ballard KJ. A comparison of two treatments for childhood apraxia of speech: methods and treatment protocol for a parallel group randomised control trial. BMC Pediatr. 2012 Aug 3;12:112. doi: 10.1186/1471-2431-12-112. PMID 22863021
- [Background] Spencer TD, Petersen DB, Adams JL. Tier 2 Language Intervention for Diverse Preschoolers: An Early-Stage Randomized Control Group Study Following an Analysis of Response to Intervention. Am J Speech Lang Pathol. 2015 Nov;24(4):619-36. doi: 10.1044/2015_AJSLP-14-0101. PMID 26125951
- [Background] Thomas DC, McCabe P, Ballard KJ. Combined clinician-parent delivery of rapid syllable transition (ReST) treatment for childhood apraxia of speech. Int J Speech Lang Pathol. 2018 Dec;20(7):683-698. doi: 10.1080/17549507.2017.1316423. Epub 2017 Apr 26. PMID 28443686